CLINICAL TRIAL: NCT01048151
Title: A PHASE I SAFETY AND TOLERABILITY TRIAL OF RADIOTHERAPY, ANDROGEN DEPRIVATION, AND INTRATUMORAL INJECTIONS OF AdGVEGR.TNF.11D (TNFeradeTM) FOR PATIENTS WITH LOCALLY ADVANCED PROSTATE CANCER
Brief Title: TNFerade Biologic to Treat Locally Advanced Prostate Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: GenVec (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Paul Fischer, PhD, CEO, GenVec
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GV-001.012
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2012-03-12 (Estimated); Status verified 2012-03

CONDITIONS: Locally Advanced Prostate Cancer
Keywords: Prostate; TNFerade Biologic
MeSH Terms: interventions — TNFeraseBiologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single (Experimental): TNFerade™ Biologic + Radiation
  Interventions: Biological: TNFerade™ Biologic

INTERVENTIONS:
Biological: TNFerade™ Biologic — AdGVEGR.TNF.11D
  Other Names: TNFerade™; AdGVEGR.TNF.11D

SUMMARY:
While radiation therapy with androgen ablation (hormone reduction) is the standard method of treating locally advanced prostate cancer. New treatments are being combined with radiation therapy in an effort to further improve the cure rates.

This study proposes to combine an experimental drug, TNFerade™ Biologic, (also called AdGVEGR.TNF.11D or "TNFerade") at different dose (amounts) levels in combination with radiation.

TNFerade™ Biologic is a form of gene transfer therapy that when injected into the tumor has shown to increase the effect of radiation therapy.

ELIGIBILITY:
Inclusion Criteria

* Histological documented high-risk localized prostate cancer defined by clinical stage >=T3 or Gleason score ≥8.
* Lack of distant metastases (including bone, liver, or extrapelvic lymph node metastases) on standard CT and bone scanning. Patients with suspected or histologically confirmed pelvic lymph node metastases are eligible.
* Normal organ function defined by:

  * Hgb > 10 mg/dl (may be transfused or on erythropoietin);
  * Platelets > 100,000/l;
  * Absolute neutrophil count > 1500/l.
* Bilirubin < 1.5 mg/dl.
* AST and ALT < 1.5X upper limit of normal.
* Written signed informed consent.

Exclusion Criteria

* Absolute or relative contraindication to prostate radiotherapy including but not limited to prior pelvic radiotherapy, active infectious or inflammatory colitis, and inability to lay supine for daily radiation treatments.
* Requirement for ongoing antithrombotic treatment with coumadin or one of its derivatives, heparin or one of its derivatives, or thrombin inhibitors. Low dose aspirin for prevention of cardiovascular events is acceptable.
* Active vascular disease defined as a stroke, transient ischemic attack (TIA), myocardial infarction, or any vascular procedure performed for ischemic disease within the last 6 months.
* History of thrombosis (pulmonary embolism (PE) or deep vein thrombosis (DVT)) or known thrombophilia.
* Coagulopathy (INR>1.5, PTT ratio >1.5)
* Major surgery within the last 1 month (excludes minor superficial surgeries, biopsies, or minimally invasive approaches).
* Chemotherapy or experimental medications within 4 weeks of study entry.
* Chronic treatment for greater than 6 months with oral steroids at doses above 10 mg/day prednisolone (or equivalent).
* Clinical evidence of active infection of any type.
* HIV-positive patients receiving combination anti-retroviral therapy.
* Other significant concurrent medical or psychiatric illness that would limit compliance with study.
* Unwilling to use condoms or another barrier method of birth control for at least 8 weeks following the last dose of TNFerade™ Biologic and some form of birth control for at least one year. -

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago, Chicago, Illinois, United States